CLINICAL TRIAL: NCT02563912
Title: Pre-calculated Doses of Medication for Pediatric Resuscitation, a Simulation Cross-over Randomized Experimental Trial
Brief Title: Pre-calculated Doses of Medication for Pediatric Resuscitation, a Simulation Experimental Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, FRCPC, St. Justine's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Resuscitaion book
Record Dates: First submitted 2015-09-27; First posted 2015-09-30 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Children; resuscitation; simulation; medication error

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handbook (Experimental): Resuscitation handbook who provides drug dosages for each weight for children. For example, at the page of 15 kg, it is written that the dosage of epinephrin is 1.5 cc of 1: 10 000.
  Interventions: Other: Handbook
- Medication chart (Active Comparator): Medication chart who provides drug dosages for each weight for children. For example,it is written that the dosage of epinephrin is 0.01 mg/kg.
  Interventions: Other: Medication chart

INTERVENTIONS:
Other: Handbook — Resuscitation handbook who provides drug dosages for each weight for children. For example, at the page of 15 kg, it is written that the dosage of epinephrin is 1.5 cc of 1: 10 000.
  Arms: Handbook
Other: Medication chart — Medication chart who provides drug dosages for each weight for children. For example,it is written that the dosage of epinephrin is 0.01 mg/kg.
  Arms: Medication chart

SUMMARY:
Dosage errors are common in the stressful situation of a pediatric resuscitation. In addition to that, studies have reported that delays to provide medication is associated to worst survival rate for very sick children. To minimize delays and error, the investigators recently published a resuscitation handbook who provides drug dosages for each weight for children thus eliminating the need for dosage calculation. Once the weight of the patient is known, the physicians only have to open the book at the page corresponding to the weight and all the medications with their calculated dosage are provided. The primary goal of this study is to evaluate the number of dosage error during simulated pediatric resuscitation comparing residents using the handbook vs. utilisation of a chart providing non-calculated dosage. This will be an experimental crossover trial among 40 residents performing four simulated case-scenarios in a high-fidelity simulation lab.

ELIGIBILITY:
Inclusion Criteria:

* Residents doing a rotation in pediatrics emergency medicine

Exclusion Criteria:

* Resident who participated in a previous month

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Having at least one dosage error in any of the medications during the case for a participant | During the simulation (10 minutes)
  Difference of > 10% of the recommended drug dosage for any of the medication provided during the simulated case scenario. To be perfect, there must be no error among all drugs provided.

SECONDARY OUTCOMES:
Dosage error in any for all individual medications during the case for a participant | During the simulation (10 minutes)
  Difference of > 10% of the recommended drug dosage for any of the medication provided during the simulated case scenario
Time for first drug prescription for each case per participant | During the simulation (10 minutes)
  Time required for the prescription of the first dose of medication. From beginning of the case until the first dose of epinephrine is completely prescribed (Dosage included)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada